CLINICAL TRIAL: NCT07014085
Title: Histomorphometric Evaluation of Bone Augmentation Using Xenograft vs Autologous Bone Graft With Dental Implants. A Comparative Clinical Study.
Brief Title: Prospective Study of Bone Augmentation With Lateral Sinus Lift and Osseointegration of Dental Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria H. Pham (Other)
Responsible Party: Sponsor-Investigator, Maria H. Pham, Associate professor, oral surgeon, DDS, PhD, University of Oslo
Organization: University of Oslo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oral surgery and Oral medicine
Record Dates: First submitted 2025-05-12; First posted 2025-06-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Atrophic Maxilla; Partial Edentulism
Keywords: bone augmentation; dento alveolar surgery; oral surgery; comparative prospective study; clinical study; lateral sinus lift; dental implants; osseointegration; prf; autologus graft; xenograft; atrophic maxilla
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Intervention Model Description: split mouth, using the participant as a control vs test group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5 years follow up study (Other): osseointegration 5 year follow up
  Interventions: Procedure: "Histomorphometric Evaluation of Bone Augmentation Using Xenografts Versus Autologous Bone Grafts in Dental Implant Patients: A Comparative Clinical Study

INTERVENTIONS:
Procedure: "Histomorphometric Evaluation of Bone Augmentation Using Xenografts Versus Autologous Bone Grafts in Dental Implant Patients: A Comparative Clinical Study — Split mouth comparative clinical prospective study xenograft vs autologous graft

SUMMARY:
By using a split-mouth model in the maxilla, lateral sinus lift procedures will be performed using xenograft on one side vs autologous bone augmentation and PRF membranes on the other side. The purpose is to qualify and verify each step of this study to ensure the reliability and validity of the results.

DETAILED DESCRIPTION:
Title: "Histomorphometric Evaluation of Bone Augmentation Using Xenografts Versus Autologous Bone Grafts in Dental Implant Patients: A Comparative Clinical Study"

Objective: This study aims to compare and analyse the effectiveness of xenograft and autologous bone grafts in bone augmentation procedures for patients requiring dental implants in a clinical setting. By comparing the outcomes of bone augmentation using xenografts and autologous bone grafts, this study aims to develop treatment protocols prioritising reduced invasiveness and enhanced efficiency. Understanding which grafting material yields better osseointegration can lead to more streamlined procedures, benefiting clinicians and patients. Furthermore, we aim to assess their efficacy in achieving optimal outcomes in bone augmentation procedures by implants and biomaterials in the study. The unique aspect of this study is the use of a split-mouth model and advanced digital technologies for data collection and analysis, which can provide more accurate and comprehensive insights into the comparative effectiveness of xenografts and autologous bone grafts.

Methodology: Utilizing a split-mouth model in the maxilla, external lateral sinus lift procedures will be performed using xenograft on one side and autologous bone augmentation and PRF membranes on the other side of the patients. A total of 20 patients will be included, with 40 implants placed. As part of the study methodology, digital technologies will be utilised for data collection and analysis. This includes digital imaging techniques for pre-operative assessment and post-operative evaluation of bone augmentation outcomes. By leveraging digital technologies, we aim to enhance the accuracy and efficiency of data collection, enabling comprehensive analysis of the comparative effectiveness of xenografts and autologous bone grafts. Rest assured, every step of this study has been meticulously planned and executed to ensure the reliability and validity of the results.

Rationale: The success of dental implants, particularly in cases of partial or total edentulism with jaw atrophy, hinges on achieving primary stability and osseointegration. Bone augmentation using either xenograft or autologous bone has been commonly employed for such treatments. However, there is an urgent need for further clinical research to evaluate the osseointegration outcomes between xenografts and autologous bone in bone augmentation procedures. The comparative analysis of xenografts and autologous bone grafts will provide crucial insights into the prevention and management of complications such as infection, graft failure, and resorption associated with bone augmentation procedures. By identifying which grafting material leads to fewer biological and technical complications, clinicians can tailor treatment protocols to minimize adverse events and maximize patient safety. This aligns with Straumann's commitment to continuously improving treatment protocols to ensure the long-term success of dental implants and restorative procedures.

Significance: With the ageing population and increasing prevalence of partial or total edentulism, the challenges associated with dental implants will continue to rise. Bone augmentation using xenografts or autologous grafts can potentially enhance implant stability and success rates, improving patients' quality of life and mental well-being. This study aims to contribute valuable insights into treatment protocols that can positively impact patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous jaws in the lateral segment with 2 or more nearby lost teeth in the posterior upper jaw (maxilla), where the vertical height is a minimum of 2mm
* absence of marginal periodontal disease
* patients in American Society of Anesthesiologists ASA group 1-2 over 18 years.

Exclusion Criteria:

* ASA group 3 and above
* ongoing infection
* bruxism or abnormal habit
* poor oral hygiene
* medical conditions that may compromise healing (uncontrolled diabetes etc)
* treatments that interfere with healing in the jaw bone (bisphosphonate, steroid therapy) radiotherapy or chemotherapy within the last 5 years
* alcohol or substance abuse
* heavy smoking
* pregnancy
* desire not to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of autogenous bone graft vs xenograft | Up to two years
  Quality measurements of bone augmentation with autologous and xenograft with histology and radiological examination
Evaluation of Bone Augmentation Using Xenografts Versus Autologous Bone Grafts Dental Implant Patients: A Comparative Clinical Study | Up til 2 years
  Measurement of survival rates and osseointegration of dental implants with questionnaires and radiology examination

SECONDARY OUTCOMES:
A prospective clinical study 3 years of follow up: Bone graft with dental implants | Up to 3 years
  Survival rate and measurements with dental implants with questionnaires and radiology examination

IPD SHARING:
Plan to Share IPD: Yes